CLINICAL TRIAL: NCT01911520
Title: Dose Finding Study for Effective Reversal of a Deep Rocuronium-induced Neuromuscular Block With Sugammadex in Morbidly Obese Patients.
Acronym: BRIDION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010/207; 2009-016857-16 (EudraCT Number)
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Morbidly Obese Patients
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- BMI < 50, Total Body Weight (TBW), 2mg/kg (Experimental): Patients with a BMI < 50, who will be dosed according to total body weight.
  Interventions: Drug: Sugammadex 2 mg/kg; Procedure: Neuromuscular monitoring.; Procedure: Clinical evaluation of residual curarization .
- BMI < 50, TBW, 4 mg/kg (Experimental): Patients with a BMI < 50, who will be dosed according to total body weight.
  Interventions: Drug: Sugammadex. 4 mg/kg; Procedure: Neuromuscular monitoring.; Procedure: Clinical evaluation of residual curarization .
- BMI < 50, Ideal Body Weight (IBW), 2 mg/kg (Experimental): Patients with a BMI < 50, who will be dosed according to ideal body weight.
  Interventions: Drug: Sugammadex 2 mg/kg; Procedure: Neuromuscular monitoring.; Procedure: Clinical evaluation of residual curarization .
- BMI < 50, IBW, 4 mg/kg (Experimental): Patients with a BMI < 50, who will be dosed according to ideal body weight.
  Interventions: Drug: Sugammadex. 4 mg/kg; Procedure: Neuromuscular monitoring.; Procedure: Clinical evaluation of residual curarization .
- BMI > 50, TBW, 2mg/kg (Experimental): Patients with a BMI > 50, who will be dosed according to total body weight.
  Interventions: Drug: Sugammadex 2 mg/kg; Procedure: Neuromuscular monitoring.; Procedure: Clinical evaluation of residual curarization .
- BMI > 50, TBW, 4mg/kg (Experimental): Patients with a BMI > 50, who will be dosed according to total body weight.
  Interventions: Drug: Sugammadex. 4 mg/kg; Procedure: Neuromuscular monitoring.; Procedure: Clinical evaluation of residual curarization .
- BMI >50, IBW, 2 mg/kg (Experimental): Patients with a BMI > 50, who will be dosed according to ideal body weight.
  Interventions: Drug: Sugammadex 2 mg/kg; Procedure: Neuromuscular monitoring.; Procedure: Clinical evaluation of residual curarization .
- BMI >50, IBW, 4 mg/kg (Experimental): Patients with a BMI > 50, who will be dosed according to ideal body weight.
  Interventions: Drug: Sugammadex. 4 mg/kg; Procedure: Neuromuscular monitoring.; Procedure: Clinical evaluation of residual curarization .

INTERVENTIONS:
Drug: Sugammadex 2 mg/kg — Patients receive 2 mg/kg Sugammadex.
  Arms: BMI < 50, Ideal Body Weight (IBW), 2 mg/kg; BMI < 50, Total Body Weight (TBW), 2mg/kg; BMI > 50, TBW, 2mg/kg; BMI >50, IBW, 2 mg/kg
Drug: Sugammadex. 4 mg/kg — Patients receive 4 mg/kg Sugammadex.
  Arms: BMI < 50, IBW, 4 mg/kg; BMI < 50, TBW, 4 mg/kg; BMI > 50, TBW, 4mg/kg; BMI >50, IBW, 4 mg/kg
Procedure: Neuromuscular monitoring. — Neuromuscular monitoring using a TOF watch SX (Organon).
Procedure: Clinical evaluation of residual curarization . — Every 30 min, during the first 2 hours after the end of the surgery.

SUMMARY:
During laparoscopic bariatric surgery, adequate muscle relaxation is important to maintain good surgical conditions. To achieve this muscle relaxation, neuromuscular transmission blocking agents, such as rocuronium (Esmeron®) are used. It sometimes happens that there is still some neuromuscular blocking activity left in the patient on awakening from anesthesia. This is called residual curarization and is known to cause postoperative complications such as impairment of respiratory function.

Sugammadex (Bridion®) is a novel drug which selectively binds rocuronium (Esmeron®). It allows for reversing of neuromuscular transmission blocking activity. Until now, all studies with sugammadex were performed in non-obese patients.

Obese patient have a high risk to suffer from post-operative respiratory failure. Therefore it is vital to avoid residual curarization. Sugammadex might be an important factor.

Obese patients have a large total body weight different from ideal body weight. Recent research demonstrated that the dose for the neuromuscular blocking agent rocuronium (Esmeron®) needs to be calculated on the patients' Ideal Body Weight rather than on Total Body Weight.

At this moment no data is available on the dose-response relationship of sugammadex in morbidly obese patients.

We hypothesize that in morbidly obese patients sugammadex should be dosed on ideal bodyweight, instead of total bodyweight.

DETAILED DESCRIPTION:
Flowchart :

72 participants

Stratification

BMI<50 BMI >50

Randomization Randomization

TBW IBW TBW IBW

2mg/kg n=9 2mg/kg n=9 2mg/kg n=9 2mg/kg n=9 4mg/kg n=9 4mg/kg n=9 4mg/kg n=9 4mg/kg n=9

TBW : Total Body Weight IBW : Ideal Body Weight

ELIGIBILITY:
Inclusion criteria :

* ASA I-II-III
* Age 18 - 65 year
* Male or female
* BMI > 30

Exclusion criteria :

* Renal failure
* Liver dysfunction
* Breastfeeding female patients, or female patients without reliable contraception
* Neuromuscular disease
* Malignant hyperthermia or a family history of malignant hyperthermia
* Allergy for neuromuscular blocking agents or other medications used during general anesthesia
* Infectious disease or patients with fever
* Patients who already received rocuronium or sugammadex on the day of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Time to complete recovery of muscle relaxation, 30 minutes after end of surgery. | 30 minutes after end of surgery.
  Measured with TOF Watch SX (TOF ratio > 0.9); clinical evaluation (eg head lift) of residual curarization in the Post Anesthetic Care.
Time to complete recovery of muscle relaxation, 1 hour after the end of surgery. | 1hour after end of surgery.
  Measured with TOF Watch SX (TOF ratio > 0.9); clinical evaluation (eg head lift) of residual curarization in the Post Anesthetic Care.
Time to complete recovery of muscle relaxation, 1 hour 30 minutes after the end of surgery. | 1hour 30 minutes after end of surgery.
  Measured with TOF Watch SX (TOF ratio > 0.9); clinical evaluation (eg head lift) of residual curarization in the Post Anesthetic Care.
Time to complete recovery of muscle relaxation, 2 hours after the end of surgery. | 2 hours after end of surgery.
  Measured with TOF Watch SX (TOF ratio > 0.9); clinical evaluation (eg head lift) of residual curarization in the Post Anesthetic Care.

SECONDARY OUTCOMES:
Need/use of rescue medication at the end of surgery | The hours following the end of surgery.
  Additional administration of sugammadex 2 mg/kg Total Body Weight) at the end of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Van Limmen, MD, Principal Investigator — University Hospital, Ghent; Luc De Baerdemaeker, MD, PhD, Principal Investigator — University Hospital, Ghent; Koen Reyntjens, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be